CLINICAL TRIAL: NCT05647187
Title: Effect Narrow-Band UVB Radiation Therapy on Suppression of IL 17 Axis in Psoriatic Patients
Brief Title: Effect Narrow-Band UVB Radiations
Acronym: UVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Hassan Mohammed Ibrahim, Associate professor of dermatology, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVU.MED.DVA021, Code 1, N76
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Psoriasis Vulgaris; UVB Phototherapy Burn
Keywords: Psoriasis vulgaris; UVB radiations; Interleukin 17

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NB-UVB group (Active Comparator): fourty patients will be treated with NB-UVB. The initial radiation dose was determined according to the patient's skin type; initial dose will be increased by 20% per session. Sessions will be given three times weekly with 48 hours apart for three months.
  Interventions: Diagnostic Test: Serum Interleukin 17 levels; Radiation: NB-UVB
- Control group (No Intervention): fourty healthy controls without psoriasis , any family history of psoriasis or any dermatological diseases.

INTERVENTIONS:
Diagnostic Test: Serum Interleukin 17 levels — Serum Interleukin 17 levels will be measured pre and post treatment by NB-UVB by performing an enzyme-linked immune sorbent assay (ELISA)
  Other Names: NB-UVB
  Arms: NB-UVB group
Radiation: NB-UVB — patients will be exposed to narrow band UVB twice weekly for three months
  Arms: NB-UVB group

SUMMARY:
Narrow-band UVR affects Interleukin 17 which has a major role in the pathogenesis of psoriasis Vulgaris. the aim of this study to evaluate the serum levels of Interleukin 17 in psoriatic patients and compare with the levels in healthy controls & evaluate the effect of narrow-band ultraviolet B (NB-UVB) on the serum of Interleukin 17 and the treatment of psoriasis Vulgaris.

DETAILED DESCRIPTION:
Nowadays Interleukin 17 has a major role in the pathogenesis of psoriasis Vulgaris.

the aim of this study to evaluate the serum levels of Interleukin 17 in psoriatic patients and compare them with the levels in healthy controls & evaluate the effect of narrow-band ultraviolet B (NB-UVB) on the serum of Interleukin 17 and the treatment of psoriasis Vulgaris. This prospective randomized clinical trial was carried out in Dermatology Department, South Valley University Hospitals included from September 2020 to August 2021, enrolled 40 psoriatic patients and 40 controls. The study was submitted for approval from the Scientific and Ethical Committees and coded as ( SVU.MED.DVA021, Code 1, N 76). Forty patients were treated with NB-UVB by starting the dose from 0.5 mJ/cm2 for all cases (Skin phototypes III or IV). The dosage is subsequently increased by 20 % per session. Sessions were given three times weekly on non-consecutive days for 12 weeks (three months). Serum Interleukin 17 levels were measured pre-and post-12 weeks narrow-band ultraviolet B by performing an enzyme-linked immune sorbent assay (ELISA). Main outcome and Measures: Improvement of psoriasis Severity Index score after 12 weeks narrow- Band UVR treatment and serum-decreased IL17 by performing an enzyme-linked immune sorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis diagnosed clinically

Exclusion Criteria:

* Patient with history of skin cancer. Patient with history of photosensitivity. Patient receiving immune suppressive drugs .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Primary (main): | 12 weeks
  To evaluate the clinical efficacy of narrow-band ultraviolet B (NB-UVB) in treatment of psoriasis vulgaris , evaluate serum levels of Interleukin 17 in psoriatic patients and compare them with levels in healthy controls

SECONDARY OUTCOMES:
Secondary (subsidiary) | 12 weeks
  Response to treatment will be evaluated by photographing the patients and calculating psoriasis area and severity index (PASI) score at the baseline before starting the treatment and monthly after starting the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Ibrahim, professor, Study Director — South Valley University
Locations (1):
- South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No